CLINICAL TRIAL: NCT03465059
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Zanubrutinib (BGB-3111) in Subjects With Varying Degrees of Hepatic Impairment
Brief Title: Safety and Pharmacokinetics of Zanubrutinib (BGB-3111) in Healthy Subjects and Those With Impaired Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-107
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Hepatic Insufficiency & Healthy Subjects
Keywords: BGB-3111; Zanubrutinib; pharmacokinetics; healthy subjects; hepatic impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Experimental): Participants with normal hepatic function will be administered a single oral dose of Zanubrutinib (80 mg).
  Interventions: Drug: Zanubrutinib
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment (Child-Pugh Class A, score of 5 to 6, inclusive) will be administered a single dose of Zanubrutinib (80 mg).
  Interventions: Drug: Zanubrutinib
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment (Child-Pugh Class B, score of 7 to 9, inclusive) will be administered a single dose of Zanubrutinib (80 mg).
  Interventions: Drug: Zanubrutinib
- Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment (Child-Pugh Class C, score of 10 to 15, inclusive) will be administered a single dose of Zanubrutinib (80 mg).
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — A single oral dose of 80 mg Zanubrutinib will be administered.

SUMMARY:
This study is designed to evaluate the safety and pharmacokinetics of zanubrutinib in subjects with impaired liver function in comparison with healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects in good health as determined by past medical history, physical examination, vital signs, ECG and laboratory tests at screening.
* Subjects must have a body mass index (BMI) between 18 and 40 kg/m2 to participate at screening.
* Female subject must be of non-childbearing potential, i.e. surgically sterile at least 6 months prior to screening with supportive clinical documentation OR post-menopausal must have no regular menstrual bleeding for at least 12 months prior to inclusion. Menopause will be confirmed by a plasma FSH level of >40 IU/L
* Male subjects must agree to practice 2 highly effective methods of birth control at least one method must be barrier technique.

Additional Inclusion Criteria for Healthy Subjects Only:

* In good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at screening; subjects without diseases/conditions
* Matched with a hepatic impaired patient (mild, moderate or severe, as applicable) using the following criteria: sex, age ±10 years and body mass index (BMI)± 10 kilograms

Additional Inclusion Criteria for Hepatic Impaired Subjects Only:

* History of cirrhosis with supportive documentation (ultrasonography, computed tomography scan, liver biopsy, magnetic resonance imaging, clinical laboratory tests results or physical signs consistent with a clinical diagnosis of liver cirrhosis.
* Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment.
* Blood pressure of 90 to 155 mmHg (systolic) and 50 to 100 mmHg (diastolic).
* Otherwise considered healthy in general as determined by physical examination findings and laboratory assessments within normal limits.

Exclusion Criteria:

* Subjects with a clinically relevant history or presence of any clinically significant disease.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* A positive human immunodeficiency virus (HIV) Type 1 or 2 test result at screening.
* History of blood donation of 500 mL or more of blood within 2 months prior to screening
* A positive tuberculosis test result.

Additional Exclusion Criteria for Hepatic Impaired Subjects Only:

* Received a liver transplant
* Acute or exacerbating hepatitis
* Active Stage 3 or 4 hepatic encephalopathy
* Previously diagnosed with hepatocellular carcinoma, or a history of cholestatic liver disease or biliary sepsis within the past 2 years.
* Additional Exclusion Criteria for Healthy Subjects Only: A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of any clinically significant chronic and/or active hepatic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Zanubrutinib (BGB-3111) to evaluate protocol specified PK parameters | Days 1, 2 & 3
  Plasma concentration of Zanubrutinib (BGB-3111) to evaluate Area Under the Plasma Concentration-Time Curve (AUC) of Zanubrutinib
Plasma concentration of Zanubrutinib (BGB-3111) to evaluate protocol specified PK parameters | Days 1, 2 & 3
  Plasma concentration of Zanubrutinib (BGB-3111) to evaluate Maximum Observed Plasma Concentration (Cmax) of Zanubrutinib

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Events (AE) | up to Day 17
  Percentage of Participants with Treatment-Emergent Adverse Events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: William Novotny, MD, Study Director — BeiGene
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ou YC, Preston RA, Marbury TC, Tang Z, Novotny W, Tawashi M, Li TK, Sahasranaman S. A phase 1, open-label, single-dose study of the pharmacokinetics of zanubrutinib in subjects with varying degrees of hepatic impairment. Leuk Lymphoma. 2020 Jun;61(6):1355-1363. doi: 10.1080/10428194.2020.1719097. Epub 2020 Feb 7. PMID 32031037